CLINICAL TRIAL: NCT00014755
Title: Phase I Pilot Study of Total-Body Irradiation, Anti-Thymocyte Globulin and Cyclophosphamide Followed By Syngeneic or Autologous Peripheral Blood Stem Cell Transplantation in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15796; FHCRC-1164.00
Record Dates: First submitted 2001-04-10; First posted 2001-04-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide; Filgrastim; Prednisone; Peripheral Blood Stem Cell Transplantation; Radiation

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: filgrastim
Drug: prednisone
Procedure: peripheral blood stem cell transplantation
Procedure: irradiation

SUMMARY:
OBJECTIVES: I. Determine the toxicity of total-body irradiation, anti-thymocyte globulin, and cyclophosphamide followed by syngeneic or autologous peripheral blood stem cell (PBSC) transplantation in patients with multiple sclerosis.

II. Determine the disease response of patients treated with this regimen. III. Determine the safety and efficacy of filgrastim (G-CSF) for PBSC mobilization in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients receive oral prednisone on days 0-10. Beginning on day 1, patients undergoing autologous peripheral blood stem cell (PBSC) transplantation receive filgrastim (G-CSF) subcutaneously daily until leukapheresis is completed. Leukapheresis begins on approximately day 4 and continues until adequate CD34+ PBSC are collected.

PBSC are collected from syngeneic donors in a similar manner. Patients undergo total-body irradiation twice daily on days -5 and -4. Patients receive cyclophosphamide IV on days -3 and -2 and anti-thymocyte globulin IV on days -5, -3, -1, 1, 3, and 5. Patients undergo autologous or syngeneic PBSC transplantation on day 0. Following PBSC transplantation, patients receive oral prednisone on days 7-30 and G-CSF IV daily beginning on day 0 and continuing until blood counts recover.

Patients are followed at 30, 80, and 90 days, monthly for 6 months, and then at 1 and 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of rapidly progressive multiple sclerosis (MS) by Proser criteria and at high risk for a fatal outcome or severe disability with one of the following:

* Primary progressive disease
* Relapsing/remitting disease with 2 or more attacks in 2 years
* Secondary progressive disease

Extended disability status scale (EDSS) between 5.0 and 8.0 with deterioration in the EDSS of 1 or more points over the past year

More than 60 days since relapse of MS

No evidence of myelodysplasia

Sibling donor proven to be an identical twin by ABO typing, HLA typing, and VNTR analysis (for syngeneic transplantation)

--Prior/Concurrent Therapy--

Radiotherapy: No prior total-lymphoid irradiation

Other: No other concurrent investigational agents

--Patient Characteristics-- Hepatic: No hepatic impairment that would preclude high-dose immunosuppressive therapy

Renal: No renal impairment that would preclude high-dose immunosuppressive therapy

Cardiovascular: No cardiac impairment that would preclude high-dose immunosuppressive therapy

Pulmonary: No pulmonary impairment that would preclude high-dose immunosuppressive therapy

Other:

* No neurologic impairment that would preclude high-dose immunosuppressive therapy
* No active uncontrolled infection
* No active malignancy
* No other illness that would severely limit life expectancy
* No medical or psychiatric conditions that would preclude study
* No history of hypersensitivity to murine proteins or E. coli-derived proteins
* No demonstrated lack of compliance with prior medical care
* Able to undergo an MRI scan
* HIV negative
* Not pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nash, Study Chair — Fred Hutchinson Cancer Center
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Bowen JD, Kraft GH, Wundes A, Guan Q, Maravilla KR, Gooley TA, McSweeney PA, Pavletic SZ, Openshaw H, Storb R, Wener M, McLaughlin BA, Henstorf GR, Nash RA. Autologous hematopoietic cell transplantation following high-dose immunosuppressive therapy for advanced multiple sclerosis: long-term results. Bone Marrow Transplant. 2012 Jul;47(7):946-51. doi: 10.1038/bmt.2011.208. Epub 2011 Nov 7. PMID 22056644